CLINICAL TRIAL: NCT04466852
Title: Otimização do Sistema de Saúde no Brasil Com Telemedicina
Brief Title: Brazilian Heart Insufficiency With Telemedicine
Acronym: BRAHIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other); University of Copenhagen (Other); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Helena DOMINGUEZ, MD, PhD, Associate Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CAAE: 14894819.5.0000.5272
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
Keywords: frail; public health; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Initial feasibility phase with patients discharged from hospital to a pilot Primary Clinic, followed by cluster randomization at Primary Clinic level, stratified by type: i. Family Clinic (with certified Family doctors) or ii. Basic Unit (mix of non-certified doctors)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardio-relay Family Clinic (Active Comparator): Patients discharged from a Rio de Janeiro municipality hospital and identified as belonging to a Family Clinic randomized to cardio-share receive instruction for telemedicine consultations. These are based on their own devices, when available, or provided by their local community agents associated in the study.
  Interventions: Other: telemedicine-guided consultation
- control Family Clinic (No Intervention): Patients discharged from a Rio de Janeiro municipality hospital and identified as belonging to a Family Clinic randomized to the control group or belonging who consent to participate in follow-up

INTERVENTIONS:
Other: telemedicine-guided consultation — Educational material is provided as short audiovisual films for understanding heart failure condition and management, how medicines work and their side effects, general advise on diets, exercise and importance of refraining from toxic exposure (smoke, alcohol, narcotics and damaging illegal medicines). Additionally, the patient (eventually assisted by their relatives and caregivers) can use this platform for learning basic important warning signs or cardiac decompensation based on feedback on recording regular measurements (weight, blood pressure and pulse and blood tests when needed) and symptoms. The cardiologist guides the patient and their Family/Basic doctors on the need for follow-up based on the parameters recorded. Videoconsultations with participation of the cardiologist, the Family/Basic doctor and the patient and relatives are used on demand.
  Arms: cardio-relay Family Clinic

SUMMARY:
A collaboration gap across sectors is a common problem in Denmark and Brazil. Brazilian Heart Insufficiency with Telemedicine (BRAHIT) will run in parallel with the ongoing Danish Reaching the Frail Elderly project (REAFEL - NCT04162548), supported by the Ministry of Higher Education and Health (Innovationsfonden - Grand Solutions), until 2021. REAFEL seeks a stronger collaboration between primary care and hospital cardiologists to manage frail elderly patients, using teleconsultation and data from mobile devices in Denmark.

Health resources are scarce in Brazil and a pressing need for the Municipal Secretary of Health of Rio de Janeiro is to reduce wait times to access some areas, as cardiology. When patients are stable after undergoing highly complex procedures in a tertiary hospital, are discharged to outpatient treatment at primary care but, a heterogenous expansion of the primary care system in the Rio de Janeiro municipality has created a great resistance from the population, and among cardiologists, to accept continuing cardiology treatment at the primary care system. Enhancing a collaboration between primary care and cardiologists, that is tangible for the patients, can relieve this pressure. The cross-sectorial collaboration in BRAHIT is based on the involvement of Instituto Nacional de Cardiologia (INC), a tertiary cardiology hospital, with primary investigator Aurora Issa (INC) and primary-and homecare in Rio de Janeiro, with primary investigator Leonardo Graever, Primary Care Special Advisor in the Municipality of Rio de Janeiro. The project proposal originates from Denmark and sponsors the project through a Danida grant (Window 2 from the Danish Foreign Ministry - Danida Fellowship Center 18-M03-KU) to the cardiologist Helena Domínguez, as associate professor in the Dept. of Biomedicine, UCPH, and consultant in Bispebjerg-Frederiksberg Hospital.

Being complex public health intervention studies, mixed methods are necessary to evaluate the value gained in the project and to provide research-based policy briefs. The methods include qualitative analyses and a cluster-randomization trial, the latter used for power calculation. Such calculation is based on adequate heart failure medications aggregated in a score constructed for this purpose. Secondary end-point is rate of number of readmissions for any cause, after discharge with heart failure diagnosis.

DETAILED DESCRIPTION:
1. AIM The aim of BRAHIT is to test a new model of care for patients with heart failure in Rio de Janeiro since the investigators can apply well-defined international guidelines for high-quality management of heart failure patients as success criteria, which have been endorsed and adapted in Brazil. Ultimately to provide a policy advice for innovative health management with telemedicine.
2. BACKGROUND Previous clinical trials that have randomized patients to conventional care or home monitoring with telemedicine solutions have failed to demonstrate a benefit of telemedicine. This is probably due to a selection bias. Accordingly, if only patients with high e-literacy, education and social level are selected for participating in telemedicine studies, it is probable that they have maximum advantage from any treatment, thus making it difficult to assess a benefit with telemedicine. In contrast, weaker patients who truly need a close care remain out of reach for cardiology expertise, remaining under primary care management, with scarce resources.

   Another problem is that, once the participants have access to the new healthcare management to be studied, conventional management gets unavoidably changed and comparison is no longer possible. Therefore, in BRAHIT, randomization will not occur at the individual patient level, but through cluster randomization at the organizational level of the primary care clinics. Successful multifaceted programs for heart failure are based on multiple visits to cardiology outpatient clinics, and patients can be safely transferred to Primary Care, but can be too strenuous for frail patients or impossible in remote areas BRAHIT includes quality indicators that allow monitoring quality of care; telemedicine-based tools for patient education, to enhance e-health literacy and innovative communication and data-exchange to support integrated care between health sectors. Telemedicine in BRAHIT can bring cardiology expertise to socially frail patients and, thereby, overcome social inequality.

   The Brazilian primary care sector is challenged with long waiting lists for referrals to specialist visits, elective surgeries, and to access higher technology services . This is aggravated in the last years, as Brazil is facing austerity measures.

   The Brazilian primary Health Care Model has evolved to almost 60% coverage, based on Family Health Teams, composed by specialized general practitioners, a nurse, nursing technicians and community health agents, while the rest are Family Health Teams with "generalists" (under-graduated physicians).

   The municipality of Rio de Janeiro, as it is particularly suitable for this project, with roughly six million habitants and a large social and cultural diversity. About 80% of the population has access to internet, electronic medical records and communication and information technology and Homecare teams are able to use social media and blogs in communicating with the local population. Therefore, it is feasible to use telemedicine communication in association with homecare teams to reach the entire population living in Rio de Janeiro. Furthermore, in BRAHIT, Primary care physicians training programs on heart failure will be based on action mapping, with adaptive technology-enhanced distance learning.
3. METHODS Participants Patients discharged from Instituto Nacional de Cardiologia (INC) with the heart failure as the primary reason for admittance (ICD-10): (DI-11.0, 13.0, 42.0, 42.6, 42.9, 50.0, 50.1, 50.9) and requests from Primary care to INC on questions for management of patients with heart failure diagnosis.

   Background population Rio de Janeiro State has nowadays 2,888 family health/homecare teams , covering 9,695,782 (57.99%) people of the State Population, and Rio de Janeiro municipality has 1.164 Family Health Teams, covering 4,016,835 people (61.61%) of the city population.

   Hypothesis A new collaboration model across sectors, using telemedicine aid, can improve the quality of care management of chronic heart disease, and reach out to weak patients. Concretely, the investigators test the hypothesis that the proportion of patients receiving correct medications for heart failure will increase from 30% to 60% in patients managed according to the BRAHIT model.

   Furthermore, the investigators hypothesize, that use of the BRAHIT model will result in a reduction of number of readmissions for heart failure within 90 days after discharge from 50% (current proportion of readmissions) to 30% (secondary end-point).

   Project design Since BRAHIT intends a complex public health intervention, it is necessary to apply mixed methods in a pragmatic manner to analyze the development and impact of the intervention. During an initial feasibility phase, unmet needs will be described based on ethnographic field observations on patients belonging to one Family Clinic that agrees to take a role as pilot-test clinic. Equivalent observations will be registered from patients discharged from INC with the selected heart failure diagnoses, who belong to other Family clinics or Basic Clinics discharged from INC Hospital.

   Patients will be informed that new procedures are being tested at INC Hospital. Data will be gathered for all patients in current clinical settings. Cluster randomization will follow with telemedicine intervention or usual care stratified by Family clinics and Basic Clinics willing to participate. Patients will be followed according to which primary care the patients belong to. The patients will be informed on what cluster their Primary Care Clinic and invited to be followed, including interviews for at least one year, until the end of the study.

   Follow-up details

   To quantify adequate use of target medications in the subgroup of patients with heart failure and reduced ejection fraction, the investigators construct a Brazilian Heart Insufficiency with Telemedicine (BRAHIT) score based on changes of clinical parameters, where higher score indicates worsening:
   * NYHA: improved or I (0 points) / no improvement (1 point) / worsening (2 points)
   * Weight: closer to target or on-target (0 points) / no change +/- 1.9 Kg since last measurement (1 point), increase 2 Kg or more (2 points)
   * ACE-I/ARB: Target dose (0 points) / tried but not reached target or not tolerated (1 point) / Never used (2 points)
   * Betablockers: Target dose (0 points) / tried but not reached target or not tolerated (1 point) / Never used (2 points)
   * Mineralocorticoid antagonist: Target dose or not indicated (0 points) / tried but not reached target or not tolerated (1 point) / Never used (2 points)

   Each patient record will have the option "unknown", when no data are available at each follow-up timepoint, to provide an indicator for data quality in the trial.

   Qualitative measurements Ethnographic observations throughout the study will be recorded and summarized at the end of the feasibility phase, identifying patient groups and elements in the process needed to reach the patients who have difficulties to receive specialized assistance when needed and an equivalent summary will be repeated based on subsequent observations until the end of the study, aiming to elucidate how use of low-cost technologies can equally reach frail and resourceful patients, regardless of the level of health literacy. Open-questions interviews will be conducted during the cluster-randomization phase to evaluate how successful the approach is from the patient perspective.

   Statistics These are a priori calculations based on expected outcomes, and they will be re-calculated based on the observations acquired during the pilot phase.

   Categorical variables will be described as absolute and relative frequencies, and continuous variables as medians (interquartile range) or means (standard deviation) according to the distribution of the variable. Normality will be evaluated with the visual inspection of histograms and application of the Shapiro-Wilks test of normality. Comparison of categorical variables will be analyzed with the Fisher exact test or chi-square for the relationship between intervention and outcomes, whereas continuous variables will be analyzed with the Mann-Whitney U test. To assess the relationship between intervention and outcomes the investigators will construct models of analysis of variance (ANOVA). These tests will be calculated as two-tailed, and p values < 0,05 will be considered significant. For evolution over time the investigators will perform Kaplan-Meier tests. The investigators use SAS, R and STATA.

   Sample size calculations for primary outcome Mortality and risk of readmission can be decreased roughly by 10% when patients are managed by multidisciplinary teams, compared to primary care management. There are no currently available data for an accurate power calculation for the population of Rio De Janeiro. Yet, based on the BREATH registry, almost 50% of the patients admitted with heart failure diagnosis are re-admitted to the hospital within 90 days after discharge, in most cases due to lack of use of relevant heart failure medications. Accordingly, 30% of patients in the cohort were admitted due to inadequate medicines for heart failure.

   Assuming a similar success to that dedicated clinics, use of beta-blockers, the most triggered treatment compliance due to side effects, can rise from less than 40% to 89% (Danish experience) or from 35 to 42% (Germany). Based on these effects, and counting on two parallel clusters, managing 26 patients in the novel collaborative BRAHIT model, there should be an improvement of adherence to the treatment from 30% to 60%, three months after discharge, with 90% power and a significance level of 5%. This shall be re-calculated with most recent data at the end of BRAHIT feasibility phase.

   Secondary outcomes In addition to the 30% admissions due to inadequate medications, many re-admissions may be due to insecurity from the primary care side. The investigators expect that the BRAHIT intervention provides a 20% absolute reduction of readmissions.
4. PUBLICATIONS AND DISSEMINATION The protocol and the results of the pilot phase of BRAHIT will be published in international peer-reviewed journals, the latter according to the extended CONSORT checklist for quantitative measurements. The findings and the evolution of the project will be described following the Template for Intervention Description and Replication (TIDieR) checklist.

Additionally, the project aims a high outreach through presentation in popular scientific media for the broader public and to publish a short policy advise that can facilitate implementation of the findings in BRAHIT.

ELIGIBILITY:
Inclusion Criteria:

* Discharge from Hospital with one of the following ICD-10 diagnoses: (DI-11.0,-13.0, 42.0, 42.6, 42.9, 50.0, 50.1, 50.9) and follow-up from INC Hospital

Exclusion Criteria:

* Patients not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
composite of all-cause mortality or at least one hospital readmission | six months after discharge
  Brasilian Heart Insufficiency with Telemedicine score based on changes in multiple parameters. For the subgroup of heart failure with reduced ejection fraction, best condition is 0 points and increasing points indicate worsening, worst 10 points and for the subgroup with preserved ejection fraction best is 0 points and worst is four points.

SECONDARY OUTCOMES:
hospital-free days | within 180 days post-discharge
  days out of hospital
serious adverse events | six months after discharge
  Based on hospital records
heart failure signs and symptoms frequency and intensity | baseline and six months after discharge
  based on patient reported outcomes
health-related quality of life | baseline and six months after discharge
  based on questionnaires (EQ-5D-5L)

OTHER OUTCOMES:
adherence to guidelines | baseline and six months after discharge
  based on electronic health records in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Helena DOMINGUEZ, MD, PhD, Study Chair — Frederiksberg hospital
Locations (2):
- Brazil (2):
  - Rio de Janeiro's Health Secretariat - Primary Care Practices, Rio de Janeiro
  - Instituto Nacional de Cardiologia Laranjeiras, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Yes
No IPD but data
Supporting Information: Study Protocol, CSR
Time Frame: Anticipated: 2 years after first inclusion - unlimited thereafter
Access Criteria: All collected IPD, all IPD that underlie results in a publication

REFERENCES:
- [Background] Bocchi EA, Marcondes-Braga FG, Bacal F, Ferraz AS, Albuquerque D, Rodrigues Dde A, Mesquita ET, Vilas-Boas F, Cruz F, Ramires F, Villacorta H Jr, Souza Neto JD, Rossi Neto JM, Moura LZ, Beck-da-Silva L, Moreira LF, Rohde LE, Montera MW, Simoes MV, Moreira Mda C, Clausell N, Bestetti R, Mourilhe-Rocha R, Mangini S, Rassi S, Ayub-Ferreira SM, Martins SM, Bordignon S, Issa VS. [Updating of the Brazilian guideline for chronic heart failure - 2012]. Arq Bras Cardiol. 2012 Jan;98(1 Suppl 1):1-33. doi: 10.1590/s0066-782x2012001000001. No abstract available. Portuguese. PMID 22392082
- [Background] Kotooka N, Kitakaze M, Nagashima K, Asaka M, Kinugasa Y, Nochioka K, Mizuno A, Nagatomo D, Mine D, Yamada Y, Kuratomi A, Okada N, Fujimatsu D, Kuwahata S, Toyoda S, Hirotani SI, Komori T, Eguchi K, Kario K, Inomata T, Sugi K, Yamamoto K, Tsutsui H, Masuyama T, Shimokawa H, Momomura SI, Seino Y, Sato Y, Inoue T, Node K; HOMES-HF study investigators. The first multicenter, randomized, controlled trial of home telemonitoring for Japanese patients with heart failure: home telemonitoring study for patients with heart failure (HOMES-HF). Heart Vessels. 2018 Aug;33(8):866-876. doi: 10.1007/s00380-018-1133-5. Epub 2018 Feb 15. PMID 29450689
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Baumann G, Honold M, Koehler K, Gelbrich G, Kirwan BA, Anker SD; Telemedical Interventional Monitoring in Heart Failure Investigators. Impact of remote telemedical management on mortality and hospitalizations in ambulatory patients with chronic heart failure: the telemedical interventional monitoring in heart failure study. Circulation. 2011 May 3;123(17):1873-80. doi: 10.1161/CIRCULATIONAHA.111.018473. Epub 2011 Mar 28. PMID 21444883
- [Background] Anker SD, Koehler F, Abraham WT. Telemedicine and remote management of patients with heart failure. Lancet. 2011 Aug 20;378(9792):731-9. doi: 10.1016/S0140-6736(11)61229-4. PMID 21856487
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835
- [Background] Niederseer D, Thaler CW, Niederseer M, Niebauer J. Mismatch between heart failure patients in clinical trials and the real world. Int J Cardiol. 2013 Oct 3;168(3):1859-65. doi: 10.1016/j.ijcard.2012.12.069. Epub 2013 Jan 25. PMID 23352093
- [Background] Thorup C, Hansen J, Gronkjaer M, Andreasen JJ, Nielsen G, Sorensen EE, Dinesen BI. Cardiac Patients' Walking Activity Determined by a Step Counter in Cardiac Telerehabilitation: Data From the Intervention Arm of a Randomized Controlled Trial. J Med Internet Res. 2016 Apr 4;18(4):e69. doi: 10.2196/jmir.5191. PMID 27044310
- [Background] Albert NM, Dinesen B, Spindler H, Southard J, Bena JF, Catz S, Kim TY, Nielsen G, Tong K, Nesbitt TS. Factors associated with telemonitoring use among patients with chronic heart failure. J Telemed Telecare. 2017 Feb;23(2):283-291. doi: 10.1177/1357633X16630444. Epub 2016 Jul 8. PMID 26869144
- [Background] Gustafsson F, Schou M, Videbaek L, Nielsen T, Ulriksen H, Markenvard J, Svendsen TL, Ryde H, Vigholt E, Hildebrandt P; Danish Heart Failure Clinics Network. Treatment with beta-blockers in nurse-led heart failure clinics: titration efficacy and predictors of failure. Eur J Heart Fail. 2007 Sep;9(9):910-6. doi: 10.1016/j.ejheart.2007.05.008. Epub 2007 Jun 14. PMID 17572146
- [Background] Schou M, Gislason G, Videbaek L, Kober L, Tuxen C, Torp-Pedersen C, Hildebrandt PR, Gustafsson F; NorthStar Investigators. Effect of extended follow-up in a specialized heart failure clinic on adherence to guideline recommended therapy: NorthStar Adherence Study. Eur J Heart Fail. 2014 Nov;16(11):1249-55. doi: 10.1002/ejhf.176. Epub 2014 Oct 14. PMID 25311554
- [Background] Schou M, Gustafsson F, Videbaek L, Tuxen C, Keller N, Handberg J, Sejr Knudsen A, Espersen G, Markenvard J, Egstrup K, Ulriksen H, Hildebrandt PR; NorthStar Investigators, all members of The Danish Heart Failure Clinics Network. Extended heart failure clinic follow-up in low-risk patients: a randomized clinical trial (NorthStar). Eur Heart J. 2013 Feb;34(6):432-42. doi: 10.1093/eurheartj/ehs235. Epub 2012 Aug 8. PMID 22875412
- [Background] Laursen DH, Frolich A, Christensen U. Patients' perception of disease and experience with type 2 diabetes patient education in Denmark. Scand J Caring Sci. 2017 Dec;31(4):1039-1047. doi: 10.1111/scs.12429. Epub 2017 May 12. PMID 28497852
- [Background] Doniec K, Dall'Alba R, King L. Austerity threatens universal health coverage in Brazil. Lancet. 2016 Aug 27;388(10047):867-8. doi: 10.1016/S0140-6736(16)31428-3. Epub 2016 Aug 25. No abstract available. PMID 27597461
- [Background] Justino AL, Oliver LL, Melo TP. Implementation of the Residency Program in Family and Community Medicine of the Rio de Janeiro Municipal Health Department, Brazil. Cien Saude Colet. 2016 May;21(5):1471-80. doi: 10.1590/1413-81232015215.04342016. English, Portuguese. PMID 27166896
- [Background] Paim J, Travassos C, Almeida C, Bahia L, Macinko J. The Brazilian health system: history, advances, and challenges. Lancet. 2011 May 21;377(9779):1778-97. doi: 10.1016/S0140-6736(11)60054-8. Epub 2011 May 9. PMID 21561655
- [Background] Soranz D, Pinto LF, Penna GO. Themes and Reform of Primary Health Care (RCAPS) in the city of Rio de Janeiro, Brazil. Cien Saude Colet. 2016 May;21(5):1327-38. doi: 10.1590/1413-81232015215.01022016. English, Portuguese. PMID 27166884
- [Background] Albuquerque DC, Neto JD, Bacal F, Rohde LE, Bernardez-Pereira S, Berwanger O, Almeida DR; Investigadores Estudo BREATHE. I Brazilian Registry of Heart Failure - Clinical Aspects, Care Quality and Hospitalization Outcomes. Arq Bras Cardiol. 2015 Jun;104(6):433-42. doi: 10.5935/abc.20150031. Epub 2015 Apr 3. PMID 26131698
- [Background] Gustafsson F, Schou M, Videbaek L, Dridi N, Ryde H, Handberg J, Hildebrandt PR; Danish Heart Failure Clinics Network. Incidence and predictors of hospitalization or death in patients managed in multidisciplinary heart failure clinics. Eur J Heart Fail. 2009 Apr;11(4):413-9. doi: 10.1093/eurjhf/hfp025. Epub 2009 Feb 21. PMID 19234309
- [Background] Gjesing A, Schou M, Torp-Pedersen C, Kober L, Gustafsson F, Hildebrandt P, Videbaek L, Wiggers H, Demant M, Charlot M, Gislason GH. Patient adherence to evidence-based pharmacotherapy in systolic heart failure and the transition of follow-up from specialized heart failure outpatient clinics to primary care. Eur J Heart Fail. 2013 Jun;15(6):671-8. doi: 10.1093/eurjhf/hft011. Epub 2013 Feb 8. PMID 23397577
- [Background] Braun V, Heintze C, Rufer V, Welke J, Stein T, Mehrhof F, Dini L. Innovative strategy for implementing chronic heart failure guidelines among family physicians in different healthcare settings in Berlin. Eur J Heart Fail. 2011 Jan;13(1):93-9. doi: 10.1093/eurjhf/hfq181. Epub 2010 Oct 14. PMID 20947573
- [Background] Campbell M, Katikireddi SV, Hoffmann T, Armstrong R, Waters E, Craig P. TIDieR-PHP: a reporting guideline for population health and policy interventions. BMJ. 2018 May 16;361:k1079. doi: 10.1136/bmj.k1079. PMID 29769210
- See also: projec description at University of Copenhagen — https://bmi.ku.dk/english/brahit